CLINICAL TRIAL: NCT01749358
Title: Optimizing the Dose of Rehabilitation After Stroke.
Brief Title: Dose Optimization for Stroke Evaluation
Acronym: DOSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Carolee Winstein, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD065438 (NIH); R01HD065438 (NIH)
Record Dates: First submitted 2012-06-25; First posted 2012-12-13 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2016-10

CONDITIONS: Stroke; Cerebrovascular Disorders; Brain Ischemia; Infarction
Keywords: stroke; hemiparesis; physical therapy; occupational therapy; neurorehabilitation; patient focused; motor learning; motor control; skill acquisition; skill training; motor recovery; task oriented training; task specific training; arm function; hand function; upper extremity; arm therapy; physical rehabilitation; arm rehabilitation; motor function
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Ischemia; Infarction; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High Therapy Dose (Experimental): Sixty total hours of ASAP therapy--challenging, intensive and meaningful practice of tasks of your choice in a collaborative partnership with your personal trainer (therapist).
  Interventions: Behavioral: Accelerated Skill Acquisition Program (ASAP)
- Moderate Therapy Dose (Experimental): Thirty total hours of ASAP therapy--challenging, intensive and meaningful practice of tasks of your choice in a collaborative partnership with your personal trainer (therapist).
  Interventions: Behavioral: Accelerated Skill Acquisition Program (ASAP)
- Low Therapy Dose (Experimental): Fifteen total hours of ASAP therapy--challenging, intensive and meaningful practice of tasks of your choice in a collaborative partnership with your personal trainer (therapist).
  Interventions: Behavioral: Accelerated Skill Acquisition Program (ASAP)
- Active Monitoring (Other): This is an observation only group.
  Interventions: Behavioral: Active Monitoring

INTERVENTIONS:
Behavioral: Accelerated Skill Acquisition Program (ASAP) — A focused, intense, evidence-based, upper extremity rehabilitation program. The training intervention is based on the fundamental elements of skill acquisition through task-specific practice, impairment mitigation to increase capacity, and motivational enhancements to build self-confidence Dosage of therapy (number of hours of therapy) will vary based on group assignment. Frequency is 4x/week, 1 week per month for 3 months in a train-wait-train paradigm. A 2-hour orientation session precedes the first visit.
  Arms: High Therapy Dose; Low Therapy Dose; Moderate Therapy Dose
Behavioral: Active Monitoring — This is an observation-only group. Any therapy received while in this group will be dosed according to usual and customary practice.
  Arms: Active Monitoring

SUMMARY:
This study is about rehabilitation of arm function after a stroke. The investigators are testing the dosage of therapy that is needed for meaningful recovery of arm and hand function. Dosage of therapy refers to the amount of time (in this case, the total number of hours) that a person participates in treatment. The investigators hope to learn how much therapy time is needed in order for change to occur in arm and hand function after a person has had a stroke. Eligible candidates must have had a stroke affecting the use of an arm or hand at least 6 months ago.

ELIGIBILITY:
Inclusion criteria:

* Ischemic or hemorrhagic stroke that occured at least 6 months ago.
* At least 21 years of age
* Persistent arm and hand weakness, with some ability to release a grasp
* Able to provide consent to participate
* No history of a medical condition that limited arm or hand use prior to the stroke
* Medically stable
* Able to participate for 10 months and attend evaluations at the University of Southern California (USC) Health Sciences Campus.
* Able to communicate in English or Spanish.

Exclusion criteria:

* Severe upper extremity sensory impairment
* Neglect
* Current major depressive disorder
* Severe arthritis or orthopedic problems that limit arm or hand movement
* Pain that interferes with daily activities
* Currently enrolled in other rehabilitation or drug intervention studies
* Living too far from the training site to participate reliably
* Receiving oral or injected anti-spasticity medications during study treatment.
* Pregnancy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Bilateral Arm Reaching Test (BART) | Change from Baseline to up to 4 months post-randomization
  BART is a laboratory-based timed-reaching task for people with stroke that was developed to evaluate upper extremity use in free-choice and forced-use scenarios. BART will be performed two times per month for the four months following randomization, and one time a month for 6 months during the follow-up period to assess changes in upper extremity use relative to dosage of therapy.
Wolf Motor Function Test (WMFT) | Change from Baseline to up to 4 months post-randomization
  Tests arm function based on time to complete 15 tasks performed with each arm. WMFT will be used to assess change in arm function relative to dose of physical therapy.
Motor Activity Log (MAL) | Change from Baseline to up to 4 months post-randomization
  Semi-structured interview in which participants are asked to rate the quality of movement (QOM) of their more affected arm for 28 activities of daily living. MAL is used to assess changes in participant perspective of arm use in daily life relative to dose of physical therapy.
Bilateral Arm Reaching Test (BART) | Change from Baseline to up to 10 months post-randomization
  BART is a laboratory-based timed-reaching task for people with stroke that was developed to evaluate upper extremity use in free-choice and forced-use scenarios. BART will be performed 2 times at Baseline, pre- and post- intervention and 1 time a month for 6 months during follow-up to assess changes in upper extremity use relative to dosage of therapy.
Wolf Motor Function Test (WMFT) | Change from Baseline to up to 10 months post-randomization
  Tests arm function based on time to complete 15 tasks performed with each arm. WMFT will be used to assess change in arm function relative to dose of physical therapy.
Motor Activity Log (MAL) | Change from Baseline to up to 10 months post-randomization
  Semi-structured interview in which participants are asked to rate the quality of movement (QOM) of their more affected arm for 28 activities of daily living. MAL is used to assess changes in participant perspective of arm use in daily life relative to dose of physical therapy.

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) | Change from Baseline to up to 4 months post-randomization
  A self-report measure to assess the ways in which an individual's health and life are impacted after a stroke. SIS will be used to assess changes in participant self-report of the impact of the stroke on health and life relative to dosage of physical therapy.
Upper Extremity Fugl-Meyer (UEFM) | Change from Baseline to up to 4 months post-randomization
  A test of motor function and sensation for the arm that is most affected by the stroke. UEFM will assess change in motor function relative to dose of physical therapy.
Stroke Impact Scale (SIS) | Change from Baseline to up to 10 months post-randomization
  A self-report measure to assess the ways in which an individual's health and life are impacted after a stroke. SIS will be used to assess changes in participant self-report of the impact of the stroke on health and life relative to dosage of physical therapy.
Upper Extremity Fugl-Meyer (UEFM) | Change from Baseline to up to 10 months post-randomization
  A test of motor function and sensation for the arm that is most affected by the stroke. UEFM will assess change in motor function relative to dose of physical therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Carolee Winstein, PhD, PT, FAPTA, Principal Investigator — University of Southern California; Nicolas Schweighofer, PhD, Principal Investigator — University of Southern California; Clarisa Martinez, PT, DPT, Study Director — University of Southern California
Locations (1):
- University of Southern California-Health Sciences Campus, Los Angeles, California, United States

REFERENCES:
- [Derived] Schweighofer N, Ye D, Luo H, D'Argenio DZ, Winstein C. Long-term forecasting of a motor outcome following rehabilitation in chronic stroke via a hierarchical bayesian dynamic model. J Neuroeng Rehabil. 2023 Jun 29;20(1):83. doi: 10.1186/s12984-023-01202-y. PMID 37386512
- [Derived] Winstein C, Kim B, Kim S, Martinez C, Schweighofer N. Dosage Matters. Stroke. 2019 Jul;50(7):1831-1837. doi: 10.1161/STROKEAHA.118.023603. Epub 2019 Jun 5. PMID 31164067